CLINICAL TRIAL: NCT06698965
Title: A Randomized, Controlled Phase II Clinical Study on the Efficacy and Safety of First-line Treatment for Extensive-stage Small Cell Lung Cancer Using a Combination Therapy of Trilaciclib, Envafolimab, Etoposide, and Carboplatin
Brief Title: Efficacy and Safety of First-line Treatment for Extensive-stage Small Cell Lung Cancer Using a Combination Therapy of Trilaciclib, Envafolimab, Etoposide, and Carboplatin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hua Zhong, Zhong Dr., MD, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS24047
Record Dates: First submitted 2024-10-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer, Small Cell
Keywords: SCLC; first-line treatment; immunotherapy; myelosuppression
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; EC regimen; envafolimab; trilaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trilaciclib+Envafolimab+Chemotherapy Group（TEC Group） (Experimental): TEC Group received received treatment with Envafolimab in combination with Etoposide and Carboplatin for 6 cycles. Prior to each chemotherapy cycle, they were given Trilaciclib before each chemotherapy session. After 6 cycles, they were treated with Trilaciclib in combination with Envafolimab as maintenance therapy until disease progression, intolerable adverse reactions, or withdrawal of informed consent by the patient occurred, with a maximum duration not exceeding 2 years.
  Interventions: Drug: Chemotherapy （Etoposide and Carboplatin）; Drug: Immunotherapy （Envafolimab）; Drug: Trilaciclib
- Envafolimab+Chemotherapy Group（EC Group） (Active Comparator): EC Group received received treatment with Envafolimab in combination with Etoposide and Carboplatin for 6 cycles. After 6 cycles, they were treated with Envafolimab as maintenance therapy until disease progression, intolerable adverse reactions, or withdrawal of informed consent by the patient occurred, with a maximum duration not exceeding 2 years.
  Interventions: Drug: Chemotherapy （Etoposide and Carboplatin）; Drug: Immunotherapy （Envafolimab）

INTERVENTIONS:
Drug: Chemotherapy （Etoposide and Carboplatin） — Etoposide: 80-100mg/m2, Q3W, intravenous infusion is administered on day 1, 2 and 3 of each cycle.
  Carboplatin: AUC=5, Q3W, intravenous infusion is administered on day 1 of each cycle.
  Other Names: Etoposide+Carboplatin
Drug: Immunotherapy （Envafolimab） — Envafolimab: 300mg, Q3W, subcutaneous injection is administered on day 1 of each cycle.
  Other Names: Envafolimab
Drug: Trilaciclib — Trilaciclib: 240mg/m2, Q3W, intravenous infusion should be completed within 4 hours before daily chemotherapy
  Arms: Trilaciclib+Envafolimab+Chemotherapy Group（TEC Group）

SUMMARY:
This prospective, randomized, controlled phase II study aims to evaluate the efficacy of combination therapy with Envafolimab and chemotherapy in first-line extensive stage SCLC, as well as the impact of Trilaciclib on the incidence of myelosuppression and anti-tumor effects in patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of gender;
* Small cell lung cancer (SCLC) confirmed by histology or cytology;
* Extensive-stage small cell lung cancer, classified as stage IV (any T, any N, M1a/b/c) according to the 8th edition of the AJCC, or T3-4 due to multiple pulmonary nodules or tumor/nodule volume too large to be included in a tolerable radiotherapy plan;
* At least one measurable lesion on imaging（RECIST 1.1）;
* Have not received any systemic anti-tumor treatment for extensive-stage diseases in the past. For patients who have received adjuvant/neoadjuvant chemotherapy in the past, or have received curative radiotherapy and chemotherapy for advanced diseases, if there is a gap of at least 6 months between disease progression or recurrence and the end of the last chemotherapy drug treatment, they are eligible to be included in this study;
* Patients with asymptomatic brain metastases or brain metastases whose symptoms have stabilized after treatment;
* Subjects are allowed to receive palliative radiation therapy (including cranial radiation therapy for symptomatic brain metastases), but the radiation therapy must be completed at least one week before enrollment;
* The laboratory test results meet the following criteria: Hemoglobin ≥ 90 g/L, neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L; Creatinine clearance rate (CrCl) ≥ 60 mL/min (as calculated using the Cockcroft-Gault formula); Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN or ≤ 5 × ULN (for patients with liver metastases); albumin ≥ 30 g/L; International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; Thyroid stimulating hormone (TSH) is within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled; The myocardial enzyme profile is within the normal range (simple laboratory abnormalities that are deemed clinically insignificant by the researchers are also allowed to be included).;
* ECOG PS score 0 or 1;
* Expected survival time ≥ 3 months;
* For Female Participants: All Female Participants with potential fertility must have a negative serum pregnancy test result during the screening period, and must take reliable contraceptive measures from signing the informed consent form until 3 months after the last dose;
* Understand and sign the informed consent form.

Exclusion Criteria:

* Diagnosed with malignant diseases other than SCLC within 5 years prior to the first administration (excluding curative basal cell carcinoma, squamous cell carcinoma, and/or excised carcinoma in situ);
* Mixed SCLC and NSCLC confirmed by histology or cytology;
* Currently participating in interventional clinical research treatment, or having received other investigational drugs or used investigational devices within 4 weeks prior to the first administration;
* Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs that stimulate or synergistically inhibit T cell receptors (such as CTLA-4, OX-40, CD137);
* Within 2 weeks before the first administration, the individual has received systematic systemic treatment with traditional Chinese patent medicines and simple preparations with anti lung cancer indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion and pleural effusion);
* Within 2 years prior to the first administration, the individual has been an active autoimmune disease requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants). Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatments;
* Within 7 days prior to the first administration of the study, the individual was receiving systemic corticosteroid therapy (excluding topical corticosteroids via nasal spray, inhalation, or other routes) or any other form of immunosuppressive therapy; Note: Physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) are allowed to be used;
* Individuals who are known to be allergic to the active ingredients or excipients of the investigational drugs, such as trilaciclib, envafolimab, etoposide, carboplatin, etc;
* Patients with clinically uncontrollable pleural/peritoneal effusion (those who do not require drainage or have no significant increase in effusion after stopping drainage for 3 days can be enrolled);
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive) or untreated active HBV, HCV;
* Pregnant or lactating female participants;
* Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA class III or IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-13 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥ 3 neutropenia during chemotherapy treatment | From enrollment to the end of Cycle 6 (each cycle is 21 days)
  According to CTCAE5.0

SECONDARY OUTCOMES:
The incidence of ≥ grade 3 thrombocytopenia or anemia during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The duration of severe neutropenia in the first treatment cycle | From enrollment to the end of Cycle 1 (each cycle is 21 days)
The incidence of febrile neutropenia during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The usage rate of granulocyte colony-stimulating factor (PEG-G-CSF/G-CSF) during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
Disease burden of patients during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
  Based on EQ-5D-5L scales scores（The score range is from 5 to 25 points, with higher scores indicating better outcomes）
The usage rate of erythropoietin (ESA) during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The usage rate of recombinant human interleukin-11 during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The usage rate of thrombopoietin (TPO) during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The usage rate of iron supplement during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The incidence of platelet transfusion during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
The incidence of red blood cell transfusion during chemotherapy | From enrollment to the end of Cycle 6 (each cycle is 21 days)
ORR | From enrollment to the end of Cycle 6 (each cycle is 21 days)
  Objective response rate
DCR | From enrollment to the end of Cycle 6 (each cycle is 21 days)
  disease control rate
DOR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Duration of response
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-Free-Survival
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  Overall survival

OTHER OUTCOMES:
Dynamic changes of immune cell subsets and cytokines in peripheral blood before and after treatment | From enrollment to the end of Cycle 6 (each cycle is 21 days)
  Including but not limited to the ratio of CD8+T/Treg and the number of T cell clones

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No